CLINICAL TRIAL: NCT01085357
Title: A Prospective, Randomized, Comparative, MultiCenter Clinical Study to Assess the Safety and Effectiveness of the Transcend CyPass Glaucoma Implant in Patients With Open Angle Glaucoma Undergoing Cataract Surgery
Brief Title: Study of an Implantable Device for Lowering Intraocular Pressure in Glaucoma Patients Undergoing Cataract Surgery
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Transcend Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMI-09-01
Record Dates: First submitted 2010-03-01; First posted 2010-03-11 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Primary Open Angle Glaucoma (POAG); Cataract
Keywords: Glaucoma; Glaucoma device; Glaucoma surgery; Intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract; Glaucoma | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CyPass Micro-Stent + Cataract Surgery (Experimental): Subjects receive the CyPass Micro-Stent at the conclusion of their cataract surgery
  Interventions: Procedure: Cataract Surgery; Device: CyPass Micro-Stent
- Cataract Surgery Only (Active Comparator): Subjects do not receive the CyPass Micro-Stent at the conclusion of their cataract surgery
  Interventions: Procedure: Cataract Surgery

INTERVENTIONS:
Procedure: Cataract Surgery — Cataract Surgery involves the removal of the natural lens, which has become clouded (called a cataract), and insertion of an artificial lens (called an intraocular lens). This procedure is done through a small surgical incision in the eye.
Device: CyPass Micro-Stent — The CyPass Micro-Stent is a small tube with a through-lumen designed to redirect aqueous fluid from the front to the back of the eye. The CyPass is implanted in the eye after completion of cataract surgery.
  Arms: CyPass Micro-Stent + Cataract Surgery

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the CyPass Implant for lowering intraocular pressure (IOP) in patients with glaucoma who undergo cataract surgery.

DETAILED DESCRIPTION:
This study is a modified and expanded protocol based on acceptable safety results from an earlier feasibility study. The trial is conducted using a 3:1 randomization (treatment to control) in which patients are screened for eligibility, randomized at time of surgery and followed for 24 months postoperatively.

ELIGIBILITY:
Preoperative Inclusion Criteria:

* Diagnosis of primary open angle glaucoma (POAG)
* Mean diurnal unmedicated IOP of 21 - 33 mmHg
* Normal anterior chamber angle anatomy at site of implantation
* Operable age-related cataract

Exclusion Criteria:

* Use of more than 3 ocular hypotensive medications (combination medications count as 2 medications)
* Significant risk associated with washout of ocular hypotensive medication
* Previous glaucoma surgery (with exception of laser treatments to the trabecular meshwork)
* Previous corneal surgery
* Clinically significant ocular pathology, other than cataract and glaucoma
* Diagnosis of acute angle closure, traumatic, congenital, malignant, uveitic, pseudoexfoliative, pigmentary or neovascular glaucoma

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 897 (Actual)
Dates: Start 2009-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President of Medical Affairs, Study Chair — Transcend Medical, Inc.

REFERENCES:
- [Derived] Ianchulev T, Lane S, Masis M, Lass JH, Benetz BA, Menegay HJ, Price FW, Lin S. Corneal Endothelial Cell Density and Morphology After Phacoemulsification in Patients With Primary Open-Angle Glaucoma and Cataracts: 2-Year Results of a Randomized Multicenter Trial. Cornea. 2019 Mar;38(3):325-331. doi: 10.1097/ICO.0000000000001826. PMID 30614901
- [Derived] Vold S, Ahmed II, Craven ER, Mattox C, Stamper R, Packer M, Brown RH, Ianchulev T; CyPass Study Group. Two-Year COMPASS Trial Results: Supraciliary Microstenting with Phacoemulsification in Patients with Open-Angle Glaucoma and Cataracts. Ophthalmology. 2016 Oct;123(10):2103-12. doi: 10.1016/j.ophtha.2016.06.032. Epub 2016 Aug 6. PMID 27506486
- [Derived] Jampel HD, Chon BH, Stamper R, Packer M, Han Y, Nguyen QH, Ianchulev T. Effectiveness of intraocular pressure-lowering medication determined by washout. JAMA Ophthalmol. 2014 Apr 1;132(4):390-5. doi: 10.1001/jamaophthalmol.2013.7677. PMID 24481483
- See also: Glaucoma Basics and Frequently Asked Questions — http://www.americanglaucomasociety.net/patients/faqs

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and randomized at 24 investigative sites located in the United States.
Pre-assignment Details: of the 897 enrolled, 392 participants were exited prior to randomization as ineligible/withdrew consent. This reporting group includes all randomized participants (505).
Groups:
- CyPass Micro-Stent + Cataract Surgery: Subjects received the CyPass Micro-Stent at the conclusion of their cataract surgery
- Cataract Surgery Only: Subjects did not receive the CyPass Micro-Stent at the conclusion of their cataract surgery
Period: Overall Study
Arm/Group | CyPass Micro-Stent + Cataract Surgery | Cataract Surgery Only
Started | 374 | 131
Completed | 355 | 125
Not Completed | 19 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Subject Decision | 4 | 3
Not completed — Investigator Decision | 1 | 1
Not completed — Death | 11 | 1
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants (Intent-to-Treat)
Groups:
- Total: Total of all reporting groups
Arm/Group | CyPass Micro-Stent + Cataract Surgery | Cataract Surgery Only | Total
Number analyzed (Participants) | 374 | 131 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (8.45) | 70.2 (8.17) | 70.3 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 72 | 269
  Male | 177 | 59 | 236

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With ≥ 20% Decrease in Intraocular Pressure (IOP) From Baseline to the Hypotensive Medication-free 24-month Postoperative Examination Using Non-responder Imputation for Missing Data
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). A reduction in IOP from baseline indicates an improvement. One eye (study eye) contributed to the analysis. Proportion of eyes is reported as a percentage. Non-responders include subject eyes for which, prior to the relevant outcome time point: 1) Use of ocular hypotensive medication was not terminated; 2) IOP-affecting secondary surgical procedure was performed; 3) CyPass was explanted; or 4) CyPass was repositioned. IOP-affecting secondary surgical procedures include: Iridotomy, iridectomy, trabeculectomy, glaucoma shunt implantation, argon laser trabeculoplasty, selective laser trabeculoplasty, or other surgery that would affect IOP. Subject eyes for which CyPass implantation was attempted but not completed were treated as non-responders.
Time Frame: Baseline; Month 24 postoperative
Population: Intent-to-treat (ITT)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | CyPass Micro-Stent + Cataract Surgery | Cataract Surgery Only
Number analyzed (Participants) | 374 | 131
Number analyzed (Eyes) | 374 | 131
percentage of eyes | 72.5 | 58.0

2. Secondary Outcome: Mean Change in IOP Between Baseline and Hypotensive Medication-free 24-month Postoperative Examination Using Baseline Value Imputation for Missing Data
Description: IOP was assessed using Goldmann applanation tonometry and reported in mmHg. A negative value indicates an improvement. One eye (study eye) contributed to the analysis. Proportion of eyes is reported as a percentage. Baseline IOP was used for subject eyes for which, prior to the relevant outcome time point: 1) Use of ocular hypotensive medication was not terminated; 2) IOP-affecting secondary surgical procedure was performed; 3) CyPass was explanted; or 4) CyPass was repositioned. IOP-affecting secondary surgical procedures include: Iridotomy, iridectomy, trabeculectomy, glaucoma shunt implantation, argon laser trabeculoplasty, selective laser trabeculoplasty, or other surgery that would affect IOP. Subject eyes for which CyPass implantation was attempted but not completed were treated as non-responders.
Time Frame: Baseline; Month 24 postoperative
Population: ITT
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CyPass Micro-Stent + Cataract Surgery | Cataract Surgery Only
Number analyzed (Participants) | 374 | 131
mmHg | -7.0 (4.53) | -5.3 (3.95)

3. Secondary Outcome: Proportion of Eyes With Postoperative IOP ≥ 6 and ≤ 18 mmHg, as Measured by Goldmann Tonometry, at the Hypotensive Medication-free 24-month Postoperative Examination Using Non-responder Imputation for Missing Data
Description: IOP was assessed using Goldmann applanation tonometry and reported in mmHg. One eye (study eye) contributed to the analysis. Proportion of eyes is reported as a percentage. Non-responders include subject eyes for which, prior to the relevant outcome time point: 1) Use of ocular hypotensive medication was not terminated; 2) IOP-affecting secondary surgical procedure was performed; 3) CyPass was explanted; or 4) CyPass was repositioned. IOP-affecting secondary surgical procedures include: Iridotomy, iridectomy, trabeculectomy, glaucoma shunt implantation, argon laser trabeculoplasty, selective laser trabeculoplasty, or other surgery that would affect IOP. Subject eyes for which CyPass implantation was attempted but not completed were treated as non-responders.
Time Frame: Month 24 postoperative
Population: ITT
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | CyPass Micro-Stent + Cataract Surgery | Cataract Surgery Only
Number analyzed (Participants) | 374 | 131
Number analyzed (Eyes) | 374 | 131
percentage of eyes | 61.2 | 43.5

ADVERSE EVENTS:
Time Frame: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury or any untoward clinical sign occurring in a study subject, whether or not related to the CyPass device. AEs were collected from time of consent to study exit (Month 24 postoperative).
Description: Reports of AEs were obtained through solicited and spontaneous comments from the subjects and through observations by the Investigator as outlined in the study protocol.
Arm/Group | CyPass Micro-Stent + Cataract Surgery | Cataract Surgery Only
Serious Adverse Events (participants affected / at risk) | 53/374 | 13/131
Other Adverse Events (participants affected / at risk) | 101/374 | 39/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CyPass Micro-Stent + Cataract Surgery (N=374) | Cataract Surgery Only (N=131)
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hiatal hernia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Biilary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Infectious colitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 2
Sepsis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Arteriogram coronary (Investigations) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Temporal lobe epilepsy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aneurysm repair (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 3 | 1
Limb operation (Surgical and medical procedures) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Knee operation (Surgical and medical procedures) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CyPass Micro-Stent + Cataract Surgery (N=374) | Cataract Surgery Only (N=131)
Worsening in visual field MD by => 2.5 dB as compared with preoperative (Nervous system disorders) | 25 | 13
AC cell and flare requiring steroid treatment at/after 30 days postoperative (Eye disorders) | 32 | 5
BCVA loss => 10 letters read at/after 3 month postoperative visit (Eye disorders) | 33 | 20
Worsening in any ocular symptom by ≥ 2 points to severe/very severe at/after 3 months postoperative (Eye disorders) | 21 | 4
Secondary ocular surgical intervention (Eye disorders) | 20 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.